CLINICAL TRIAL: NCT04388163
Title: Effects of Gentian Violet Treatment on Patients With Hidradenitis Suppurativa
Brief Title: Gentian Violet Treatment for Hidradenitis Suppurativa
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug company did not approve use of the drug, IRB never approved
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00063737
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hidradenitis Suppurativa
Keywords: HS; Gentian Violet; nonsurgical treatment
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Gentian Violet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gentian Violet Treatment (Experimental): A single application of gentian violet will be topically applied to the site(s) of active HS involvement by a trained staff member. The sites will then be bandaged by staff and patients will be instructed about home maintenance procedures.
  Interventions: Drug: Gentian Violet

INTERVENTIONS:
Drug: Gentian Violet — Gentian violet is a topical antiseptic used to treat many cutaneous yeast infections. It also has a role in improving wound healing in sites of active ulceration.
  Other Names: crystal violet

SUMMARY:
This is a survey study being conducted to describe how subjects with Hidradenitis suppurativa (HS) respond to treatment with gentian violet. The study will rely primarily on qualitative survey responses and quantitative changes in skin appearance.

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is a chronic disease of the folliculopilosebaceous unit, often found in intertriginous areas of the body. The pain and impairment of HS leads patients to report a decreased quality of life, even in comparison to other debilitating cutaneous disease states. Pharmalogic management of HS can vary from topical antibiotics or intralesional corticosteroids for mild cases to immunosuppressants and biologic agents in refractory cases. Gentian violet is a topical antiseptic used to treat many cutaneous yeast infections. It also has a role in improving wound healing in sites of active ulceration. It is our hypothesis that gentian violet will help minimize skin trauma in sites of active HS to promote improved wound healing and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have active HS, be willing to undergo one application of HS, and agree to follow-up in one month.

Exclusion Criteria:

* Exclusion criteria include children, absent HS lesions at the time of clinic, and cognitive/physical impairments that would make them unable to assess quality of life factors of the survey.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Skin's Redness | baseline pre-treatment
  Subjects rate site redness on a scale from 1 (no redness) to 5 (severe redness)
Skin's Redness | 1 month post-treatment
  Subjects rate skin redness at treatment site on a scale from 1 (no redness) to 5 (severe redness)
Skin's Drainage | baseline pre-treatment
  Subjects rate skin drainage at treatment site on a scale from 1 (no drainage) to 5 (severe drainage)
Skin's Drainage | 1 month post-treatment
  Subjects rate skin drainage at treatment site on a scale from 1 (no drainage) to 5 (severe drainage)
Skin's Pain | baseline pre-treatment
  Subjects rate skin pain at treatment site on a scale from 1 (no pain) to 5 (severe pain)
Skin's Pain | 1 month post-treatment
  Subjects rate skin pain at treatment site on a scale from 1 (no pain) to 5 (severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Pichardo-Geisinger, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No